CLINICAL TRIAL: NCT07134153
Title: Evaluating Safety and Efficacy of INtrathecal or Ommaya ReserVoir Administration of T-DXd in Patients With HER2-Expressing Breast Cancer With Active Leptomeningeal and/or Brain Metastases Based on Systemic Therapy: Phase I/II Study
Brief Title: Phase I/II Study of Intrathecal/Ommaya T-DXd in HER2-Expressing Breast Cancer With Leptomeningeal/Brain Metastases
Acronym: INOVATE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Director of Phase I Clinical Trial Department; Professor, Chief physician of oncology department, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2501313-7
Record Dates: First submitted 2025-05-11; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Phase I/Arm A(Intrathecal Dose-Escalation Phase) (Experimental): Population : T-DXd-naïve subjects with leptomeningeal metastases (LM), with or without concurrent brain metastases (BM).
  Cycle 1 : Intrathecal (IT) T-DXd monotherapy to assess cerebrospinal fluid (CSF) and systemic pharmacokinetics (PK).
  Cycles 2+ : IT T-DXd combined with intravenous (IV) T-DXd in a dose-escalation design to determine the maximum tolerated dose (MTD) .
  DLT Evaluation : The first two cycles serve as the dose-limiting toxicity (DLT) observation window .
  Endpoint : The recommended Phase 2 dose (RP2D) will be determined by investigator assessment
  Interventions: Drug: T-DXd
- Phase I/Arm B(Systemic-to-Intrathecal Transition Phase) (Experimental): Population : T-DXd-naïve subjects with LM ± BM. Cycle 1 : IV T-DXd monotherapy to characterize CSF and systemic PK profiles. Cycles 2+ : IT administration of the RP2D of T-DXd combined with IV therapy
  Interventions: Drug: T-DXd
- Phase II/Arm A (Experimental): HER2-positive advanced breast cancer with progressive leptomeningeal and/or brain metastases after prior T-DXd therapy
  Interventions: Drug: T-DXd
- Phase II/Arm B (Experimental): HER2-low (IHC 1+ or 2+/ISH-) advanced breast cancer with progressive leptomeningeal and/or brain metastases after prior T-DXd therapy
  Interventions: Drug: T-DXd
- Phase II/Arm C (Experimental): HER2-positive advanced breast cancer with progressive brain metastases (without leptomeningeal involvement) after prior T-DXd therapy
  Interventions: Drug: T-DXd
- Phase II/Arm D (Experimental): HER2-low advanced breast cancer with progressive brain metastases (without leptomeningeal involvement) after prior T-DXd therapy
  Interventions: Drug: T-DXd
- Phase II/Arm E (Experimental): T-DXd-naïve HER2-positive advanced breast cancer with progressive leptomeningeal and/or brain metastases
  Interventions: Drug: T-DXd
- Phase II/Arm F (Experimental): T-DXd-naïve HER2-low advanced breast cancer with progressive leptomeningeal and/or brain metastases
  Interventions: Drug: T-DXd
- Phase II/Arm G (Experimental): T-DXd-naïve HER2-positive advanced breast cancer with progressive brain metastases (without leptomeningeal involvement)
  Interventions: Drug: T-DXd
- Phase II/Arm H (Experimental): T-DXd-naïve HER2-low advanced breast cancer with progressive brain metastases (without leptomeningeal involvement)
  Interventions: Drug: T-DXd

INTERVENTIONS:
Drug: T-DXd — Evaluating safety and efficacy of intrathecal or ommaya reservoir administration of T-DXd in patients with HER2-expressing breast cancer with active leptomeningeal and/or brain metastases based on systemic therapy
  Other Names: DS8201a

SUMMARY:
Multiple trials confirm systemic T-DXd efficacy in HER2+ breast cancer with leptomeningeal/brain metastases, yet median LM survival remains 3-4 months, highlighting unmet needs. While systemic therapies improve survival, intracranial disease control remains limited due to poor BBB penetration. Preclinical data show no detectable T-DXd/DXd in CSF, though intrathecal trastuzumab demonstrates preliminary safety/efficacy in HER2+ LM.

This study evaluates intrathecal/intra-Ommaya T-DXd plus systemic therapy in active HER2+ meningeal/brain metastases, assessing safety, intracranial efficacy, and CSF/peripheral blood T-DXd distribution to clarify BBB penetration potential. Findings may guide novel therapeutic strategies for this high-need population.

DETAILED DESCRIPTION:
Multiple clinical trials have demonstrated the efficacy of systemic T-DXd in advanced HER2-expressing breast cancer with leptomeningeal and/or brain metastases. However, the median survival of leptomeningeal metastasis (LM) patients remains only 3-4 months, and treatment options for isolated brain metastases are limited, underscoring the need for more effective therapeutic strategies.

While systemic therapies have prolonged survival in advanced breast cancer, intracranial disease management remains constrained by a lack of effective local treatments. As the use of T-DXd increases, the progression of intracranial lesions in patients who have received prior local therapy or lack indications for radiotherapy has become a critical unmet clinical challenge.

Conventional understanding holds that large biologic molecules poorly penetrate the blood-brain barrier (BBB). Preclinical studies detected neither T-DXd nor free DXd (payload) in cerebrospinal fluid (CSF), and the distribution of T-DXd in human CSF remains uncharacterized. However, preliminary data suggest that intrathecal trastuzumab-alone or combined with pertuzumab-exhibits acceptable safety and efficacy in HER2-positive LM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, regardless of gender.
* HER2-expressing advanced or metastatic breast cancer
* Leptomeningeal metastasis
* Subjects with active brain metastases only must have at least one intracranially measurable lesion (RANO-BM criteria).
* Adequate organ and bone marrow function
* No radiotherapy, chemotherapy, targeted therapy, immunotherapy, endocrine therapy, or surgery within 2 weeks prior to enrollment (or within 5 half-lives of prior therapy, whichever is shorter).
* All prior treatment-related toxicities must have resolved to ≤Grade 1

Exclusion Criteria:

* Diagnosis of other malignancies within the past 5 years, except for cured carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin, other in situ carcinomas, or papillary thyroid carcinoma.
* Uncontrolled concurrent illnesses including, but not limited to: persistent or active infections, uncontrolled or clinically significant cardiovascular diseases, severe chronic gastrointestinal disorders with diarrhea, or psychiatric/social conditions that may compromise compliance with study requirements, significantly increase AE risks, or impair the subject's ability to provide written informed consent.
* History of (non-infectious) ILD/non-infectious pneumonitis requiring steroid therapy, current ILD/non-infectious pneumonitis, or suspected ILD/non-infectious pneumonitis that cannot be ruled out by imaging during screening.
* Clinically significant pulmonary comorbidities
* Use of immunosuppressants or systemic corticosteroids (>10 mg/day prednisone equivalent) for immunosuppression within 2 weeks prior to first dose (excluding intranasal/inhaled corticosteroids).
* Any active autoimmune disease or history of autoimmune disease with potential recurrence.
* Uncontrolled infections requiring IV antibiotics, antivirals, or antifungals.
* Active primary immunodeficiency, known HIV infection, active HBV (HBsAg+ with HBV DNA ≥500 IU/mL) or HCV infection. HCV antibody-positive subjects are eligible only if PCR confirms HCV RNA negativity.
* Radiographic evidence of tumor encasement/invasion of major blood vessels, or investigator-determined high risk of fatal hemorrhage due to probable vascular invasion during treatment.
* Pregnant/lactating women, or subjects of reproductive potential unwilling/unable to use effective contraception.
* Any other condition deemed by investigators to potentially affect trial conduct or outcome interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Phase I Stage Cohort A: Maximum Tolerated Dose (MTD) | Up to 21 days after the first dose
  Cohort A: Maximum Tolerated Dose (MTD) of intracapsular administration，In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Phase I Stage Cohort B: Maximum serum concentration (Cmax) | Up to 21 days after the first dose
  Cohort B: Maximum serum concentration (Cmax) of T-DXd in cerebrospinal fluid and blood will be investigated.
Phase I Stage Cohort B:Time to maximum serum concentration (Tmax) | Up to 21 days after the first dose
  Cohort B: Time to maximum serum concentration (Tmax) of T-DXd in cerebrospinal fluid and blood will be investigated.
Phase I Stage Cohort B:Half-life (T1/2) | Up to 21 days after the first dose
  Cohort B: Half-life (T1/2) of T-DXd in cerebrospinal fluid and blood will be investigated.
Phase II Stage Cohorts A: LM-OS | 18 months
  Cohorts A: leptomeningeal metastasis-overall survival（LM-OS）
Phase II Stage Cohorts B: LM-OS | 18 months
  Cohorts B: leptomeningeal metastasis-overall survival（LM-OS）
Phase II Stage Cohorts C: LM-ORR | 18 months
  Cohorts C: leptomeningeal metastasis-Objective Response Rate（LM-ORR）
Phase II Stage Cohorts D: LM-ORR | 18 months
  Cohorts D: leptomeningeal metastasis-Objective Response Rate（LM-ORR）
Phase II Stage Cohorts E: LM-OS | 18 months
  Cohorts E: leptomeningeal metastasis-overall survival（LM-OS）
Phase II Stage Cohorts F: LM-OS | 18 months
  Cohorts F: leptomeningeal metastasis-overall survival（LM-OS）
Phase II Stage Cohorts G: LM-ORR | 18 months
  Cohorts G: leptomeningeal metastasis-Objective Response Rate（LM-ORR）
Phase II Stage Cohorts H: LM-ORR | 18 months
  Cohorts H: leptomeningeal metastasis-Objective Response Rate（LM-ORR）

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Cancer, Shanghai, Shanghai Municipality